CLINICAL TRIAL: NCT04851496
Title: A Study to Evaluate the Ability of Speech- and Language-based Digital Biomarkers to Detect and Characterise Prodromal and Preclinical Alzheimer's Disease in a Clinical Setting - PAST Extension Study.
Brief Title: Amyloid Prediction in Early Stage Alzheimer's Disease From Acoustic and Linguistic Patterns of Speech - PAST Extension
Acronym: AMYPRED-PAST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Novoic Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: NOV-0100-2
Record Dates: First submitted 2021-04-12; First posted 2021-04-20 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2021-04

CONDITIONS: Alzheimer Disease; Preclinical Alzheimer's Disease; Prodromal Alzheimer's Disease; Alzheimer's Disease (Incl Subtypes); Mild Cognitive Impairment
Keywords: Alzheimer's disease; Preclinical Alzheimer's disease; Prodromal Alzheimer's disease; Mild Cognitive Impairment; Normal Cognition; Amyloid; Speech; Acoustic; Language; Linguistic; Machine Learning; Artificial Intelligence
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Speech; Language

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Arm 1: MCI amyloid positive: * Meet the National Institute of Aging - Alzheimer's Association (NIA-AA) core clinical criteria (2011) for MCI due to Alzheimer's or Mild Alzheimer's Dementia
  * Positive amyloid PET or amyloid CSF status.
  * MMSE 23-30 (inclusive)
- Arm 2: MCI amyloid negative: * Non-AD Mild Cognitive Impairment (MCI)
  * Negative amyloid PET or amyloid CSF status.
  * MMSE 23-30 (inclusive)
- Arm 3: CN amyloid positive: * Absence of a diagnosis of cognitive disorder and/or subjectively reported cognitive decline
  * Positive amyloid PET or amyloid CSF status.
  * MMSE 26-30 (inclusive)
- Arm 4: CN amyloid negative: * Absence of a diagnosis of cognitive disorder and/or subjectively reported cognitive decline
  * Negative amyloid PET or amyloid CSF status.
  * MMSE 26-30 (inclusive)

SUMMARY:
The primary objective of the study is to evaluate whether a set of algorithms analysing acoustic and linguistic patterns of speech can detect amyloid-specific cognitive impairment in early stage Alzheimer's disease, based on archival spoken or written language samples, as measured by the AUC of the receiver operating characteristic curve of the binary classifier distinguishing between amyloid positive and amyloid negative arms. Secondary objectives include (1) evaluating how many years before diagnosis of MCI such algorithms work, as measured on binary classifier performance of the classifiers trained to classify MCI vs cognitively normal (CN) arms using archival material from the following time bins before MCI diagnosis: 0-5 years, 5-10 years, 10-15 years, 15-20 years, 20-25 years; (2) evaluating at what age such algorithms can detect later amyloid positivity, as measured on binary classifier performance of the classifiers trained to classify amyloid positive vs amyloid negative arms using archival material from the following age bins: younger than 50, 50-55, 55-60, 65-70, 70-75 years old.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are fully eligible for and have completed the AMYPRED (Amyloid Prediction in early stage Alzheimer's disease from acoustic and linguistic patterns of speech) study.

(See https://clinicaltrials.gov/ct2/show/NCT04828122)

* Subject has access to audio or written recordings created by them that are available for collection.
* Subject consents to take part in PAST extension study.

Exclusion Criteria:

* Subject hasn't completed the full visit day in the AMYPRED study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be identified from participants of the AMYPRED study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is the area under the curve (AUC) of the receiver operating characteristic (ROC) curve of the binary classifier distinguishing between amyloid positive (Arms 1 and 3) and amyloid negative (Arms 2 and 4) arms. | Up to 85 years
  Using archival spoken or written language samples as input.

SECONDARY OUTCOMES:
The sensitivity, specificity and Cohen's kappa of the binary classifier distinguishing between amyloid positive (Arms 1 and 3) and amyloid negative (Arms 2 and 4) arms using archival spoken or written language samples as input. | Up to 85 years
The AUC, sensitivity, specificity and Cohen's kappa of the binary classifiers distinguishing between MCI and cognitively normal (CN) arms. | Up to 85 years
  Using archival spoken or written language samples as input in the following bins: 0-5 years, 5-10 years, 10-15 years, 15-20 years, 20-25 years before MCI diagnosis.
The AUC, sensitivity, specificity and Cohen's kappa of the binary classifier distinguishing between amyloid positive (Arms 1 and 3) and amyloid negative (Arms 2 and 4) arms. | Up to 85 years
  Using archival spoken or written language samples as input in the following bins: younger than 50, 50-55, 55-60, 65-70, 70-75 years old.

CONTACTS AND LOCATIONS:
Overall Officials: Emil Fristed, MSc, Principal Investigator — Novoic Limited
Locations (4):
- United Kingdom (4):
  - Re:Cognition Health, Birmingham
  - Re:Cognition Health, Guildford
  - Re:Cognition Health, London
  - Re:Cognition Health, Plymouth

IPD SHARING:
Plan to Share IPD: Undecided